CLINICAL TRIAL: NCT04845464
Title: The Relationship Between Sleep Quality and Cognition in Young Adults
Brief Title: Sleep Quality and Cognition in Young Adults
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, mbudak, Asst. Prof. Miray Budak. Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: SleepCog2021
Record Dates: First submitted 2021-04-10; First posted 2021-04-15 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Healthy Adults
Keywords: Sleep Quality; Cognitive Status; healthy adult
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: A group of young adults aged between 18 to 25
  Interventions: Other: Cognitive Assessment (not diagnostic)

INTERVENTIONS:
Other: Cognitive Assessment (not diagnostic) — Sleep quality and cognition will be assessed in young adults

SUMMARY:
Sleep quality is impaired in young adults due to current conditions. Recent studies emphasize that this situation may also affect the cognitive status of individuals. The aim of this study was to investigate the relationship between sleep quality and cognitive status in young adults. A total of 122 young adults (61 female, 61 male) aged between 18 to 25 and studied at Istanbul Medipol University, Faculty of Health Sciences, were included in the study. Individuals were evaluated with "Pittsburgh Sleep Quality Index (PSQI)" for sleep quality; with "Montreal Cognitive Status Scale (MoCA)" for cognitive status, with "STROOP Test" for selective attention; with "Verbal Fluency Test" for sustained attention; with "WMS-R digit Span Test" for auditory attention

ELIGIBILITY:
Inclusion Criteria:

* Signing the Informed Voluntary Consent Form
* Being in the age range of 18-25

Exclusion Criteria:

* having a sleep disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults aged between 18 to 25
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 8 March - 26 April 2019
  Pittsburgh Sleep Quality Index evaluates sleep quality and impairment in the last one month. 19 of the 24 PSQIquestions included were self-report questions. The scale has 18 questions and 7 components: Subjective Sleep Quality "," Sleep Latency "," Sleep Duration ", "Sleep Efficiency", "Sleep Disturbance", "Sleep Medication" and Daytime Dysfunction". The total score ranges from 0-21. A total score greater than 5 indicates poor sleep quality.
Montreal Cognitive Assessment Test | 8 March - 26 April 2019
  Montreal Cognitive Assessment Test (MoCA) examines cognitive abilities such as visual / executive function, naming, episodic memory, attention, language, abstract thinking, and orientation. The original cut-off score of the MoCA test is 26. The cut-off score of 21 was adopted in Turkey. MoCA takes about 10 minutes to apply, but shortened versions have been created to shorten the administration time

SECONDARY OUTCOMES:
STROOP Test | 8 March - 26 April 2019
  The Stroop Test reflects selective attention, reading and color rendering processes. It is a critical experimental task, often used in the study of automatic and parallel processing models with the speed of information processing. Because of these features, the test is used not only in the evaluation of the cognitive processes of healthy individuals, but also in the evaluation of many psychiatric and neurological disorders
Verbal Fluency Test | 8 March - 26 April 2019
  Verbal Fluency Test evaluates the tasks performed with frontal and temporal lobe activation. The purpose of this test is to evaluate the mental recall of words starting with the given letter or in the desired category within the prescribed time.
WMS-R digit Span Test | 8 March - 26 April 2019
  Digit Span Test is the eighth subtest in the Wechsler Memory Scale Developed Form, and evaluates the simple and complex attention of individuals. This sub-test consists of two sub-sections, and a series of increasingly long numbers are read to the person. Both subtests are related to auditory attention and short-term memory. Two separate trials are made for each length sequence.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No